CLINICAL TRIAL: NCT04646057
Title: The Safety and Effectiveness of DuraSorb® for Reinforcement in Patients Undergoing Prosthetic Breast Reconstruction
Brief Title: DuraSorb® in Prosthetic Breast Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Surgical Innovation Associates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-004
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2023-11

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment Arm (Experimental)
  Interventions: Device: DuraSorb®
- Historical Control Arm (No Intervention)

INTERVENTIONS:
Device: DuraSorb® — Monofilament Surgical Mesh
  Arms: Treatment Arm

SUMMARY:
This study compares outcomes of prospective mesh-based breast reconstructions to historical control breast reconstructions with no mesh.

DETAILED DESCRIPTION:
Plastic surgeons have a variety of biologic and synthetic mesh available for use. However, no mesh has adequately evaluated safety and effectiveness for FDA approval or clearance for use in breast reconstruction. Therefore, no mesh is an appropriate comparator for a randomized clinical study.

This multi-center, prospective, clinical study with matched historical controls of total submuscular 2-stage breast reconstructions with no mesh will evaluate the safety and effectiveness of DuraSorb® monofilament surgical mesh when implanted in subjects undergoing 2-stage breast reconstruction.

Women scheduled for mastectomy and immediate 2-stage breast reconstruction will sign informed consent and satisfy eligibility criteria prior to the first stage of surgery and DuraSorb® implantation.

Maximum study follow-up is through one year after definitive reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Female between the inclusive ages of 22 and 70 at the time of initial expander surgery
* Scheduled to undergo either unilateral or bilateral mastectomy with immediate 2-stage breast reconstruction
* Is able to understand the study requirements and is willing to provide written informed consent
* Is willing and able to return for all scheduled study visits

Exclusion Criteria:

* Is pregnant or planning to become pregnant during study participation
* Has a history of failed tissue expansion or breast implantation at the intended reconstruction site
* has a residual gross tumor at the intended reconstruction site
* has been treated for a systemic infection or a local infection at the surgical site that the investigator determines will affect the safety of the subject during breast reconstruction and/or mesh use
* has, as determined by the investigator, unsuitable tissue integrity for immediate 2-stage breast reconstruction
* has undergone previous radiation therapy to the reconstruction site or chest wall
* is scheduled to undergo post-operative radiation therapy at the reconstruction site
* has a Body Mass Index (BMI) < 14 or > 44
* has used nicotine products within 90 days of screening
* is currently taking medications including non-NSAID anti-coagulants, immunosuppressants (including systemic steroids), or other medications determined by the investigator to place the subject at an increased risk of local complications of breast reconstruction
* has been diagnosed with a comorbid condition determined by the investigator to place the subject at an increased risk of complications
* has participated in any other clinical study that the investigator feels may interfere with this clinical study

Ages: 22 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Composite Clinical Success (CCS) | 12 Month Follow-Up
  This outcome measure is a combination of effectiveness and safety components. CCS is defined as intraoperative fill volume of at least 45% of the total expander size and the absence of expander or implant removal for cause or major cosmetic revision between the DuraSorb Treatment Arm and historical controls.
Local Complications of Breast Reconstruction | 12 Month Follow-Up
  The rates of a set of breast reconstruction complications (i.e. infection, serum, necrosis, etc.) will be measured between the DuraSorb Treatment Arm and historical controls.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Northwestern Specialists Plastic Surgery, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Harvard Brigham and Women's Faulkner Hospital, Boston, Massachusetts
  - NYU Grossman School of Medicine, New York, New York
  - Kelsey-Seybold Clinic, Houston, Texas
  - University of Wisconsin Health University Hospital, Madison, Wisconsin